CLINICAL TRIAL: NCT07056504
Title: Active Rehabilitation Training System for Motor and Cognitive Function Technologies and Systems for Assessing Human Energy Metabolism and Nutritional Rehabilitation
Brief Title: Technologies and Systems for Assessing Human Energy Metabolism and Nutritional Rehabilitation
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Xueying Zhang, Principal investigator, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-250615-H0986
Record Dates: First submitted 2025-06-17; First posted 2025-07-09 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Energy Metabolism; Nutrition, Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will collect patients' urine samples to measure energy expenditure, blood samples for metabolomics and hormone level analysis, and fecal samples for microbiome profiling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rehabilitation: Individuals aged 20 to 70 years, who are recovering from stroke or motor injuries

SUMMARY:
The objective of this observational study is to integrate the doubly labeled water (DLW) database from healthy individuals with multimodal data-including, but not limited to, weight, height, age, sex, race, elevation-from cohorts undergoing rehabilitation following movement impairments or neurological injuries. Machine learning algorithms will be used to develop injury-specific predictive models of energy requirements.

The primary research question is:

How does energy metabolism change during the rehabilitation process in individuals recovering from traumatic brain injury, stroke, or major surgical procedures? To answer this, participants will undergo a comprehensive set of assessments, including measurements of height and weight, body composition, resting metabolic rate, physical activity levels, total energy expenditure, psychological health, food intake and hunger ratings, sleep quality, cognitive performance, non-invasive brain function monitoring, and gait analysis. Fecal and blood samples will also be collected for untargeted metabolomics analysis.

DETAILED DESCRIPTION:
1. Body Weight and Height Participants will fast overnight prior to measurement. Body weight will be measured in the morning using a calibrated Seca digital scale, with participants wearing light clothing and no shoes. Height will be measured using a Seca 217 stadiometer, with participants standing barefoot.
2. Resting Energy Expenditure (REE) REE will be measured via indirect calorimetry using a respiratory hood system (Cosmed). Participants will report to the laboratory after an overnight fast, lie supine on a flat bed, and have the hood placed over their head. Oxygen consumption and carbon dioxide production will be recorded for 40 minutes, with the final 10 minutes used for analysis. The system will be quality-checked regularly using a turbine test, and monthly validation will be conducted via an alcohol combustion test.
3. Total Energy Expenditure (TEE)

   TEE will be assessed using two complementary methods:

   Doubly Labeled Water (DLW) Method: Urine samples from the DLW subset will be stored at -20 °C and shipped on dry ice to Shenzhen Institutes of Advanced Technology, Chinese Academy of Sciences. Isotope ratios will be analyzed using a Liquid Water Isotope Analyzer (ABB). CO₂ production will be calculated using the latest equation from Speakman et al. (2021, Cell Reports Medicine), and TEE will be estimated using the Weir equation.

   Metabolic Chamber: TEE will also be measured using a whole-body metabolic chamber (Maastricht Instruments, Netherlands), which continuously tracks oxygen consumption and carbon dioxide production. Participants will remain in the chamber for 48 hours, engaging in routine daily activities. Data from the second day will be analyzed to estimate TEE.
4. Physical Activity Physical activity will be assessed using a GT3X accelerometer worn on the hip for 15 consecutive days. The device should not be worn during bathing or swimming. Data from the first day and any day with <12 hours of wear time will be excluded. A valid dataset requires at least two weekdays and two weekend days of usable data.
5. Body Composition

   Body composition will be measured using the following techniques:

   Magnetic Resonance Imaging (MRI; Philips Multiva 1.5T) Dual-energy X-ray Absorptiometry (DXA; HOLOGIC Horizon Wi, USA) Bioelectrical Impedance Analysis (BIA; TANITA MC-980, Japan) Parameters to be assessed include total and regional fat mass, lean mass, and fat percentage across the limbs and trunk. MRI will be used for whole-body fat distribution analysis by trained technicians.
6. Mental Health Assessment The Symptom Checklist-90 (SCL-90) will be used to evaluate psychological well-being. This tool measures ten dimensions: somatization, obsessive-compulsive traits, interpersonal sensitivity, depression, anxiety, hostility, phobia, paranoid ideation, psychosis, and additional symptoms. Scores for each dimension and overall symptom severity will be calculated.
7. Food Intake and Hunger Assessment Meals will be designed based on the energy distribution guidelines from the Chinese Dietary Guidelines. After a standardized lunch, participants will receive a test meal (packaging removed) containing predefined macronutrient and energy levels five hours later. Food intake will be ad libitum, and hunger levels will be assessed based on behavioral indicators. Blood samples (4 mL) will be collected at baseline (pre-dinner), and 15, 30, and 60 minutes post-dinner for appetite-related hormones analysis such as ghrelin and PYY.
8. Sleep Quality Monitoring Sleep will be monitored using the Heartcare Youhu Pro AI Precision Health Management System, which tracks total sleep duration, sleep efficiency, cycle durations, heart rate, and respiratory patterns. These metrics will be used to assess sleep quality.
9. Cognitive Function Assessment

   Cognitive performance will be evaluated using:

   Mini-Mental State Examination (MMSE): Assesses orientation, memory, attention, language, and visuospatial function. Scores of 25-30 indicate normal function; 20-24 mild, 10-19 moderate, and <10 severe cognitive impairment.

   Montreal Cognitive Assessment (MoCA): Screens for impairment across eight cognitive domains. A score ≥26 is considered normal.
10. Non-Invasive Brain Function Monitoring Functional Near-Infrared Spectroscopy (fNIRS) will be used to assess brain activity by measuring changes in oxyhemoglobin and deoxyhemoglobin concentrations. We may use the BS2000 near-infrared imaging system for this purpose.

    Assessment Areas: Prefrontal cortex, motor cortex, frontal pole, dorsolateral prefrontal cortex, primary motor/somatosensory cortex, premotor and supplementary motor cortex-on both healthy and affected sides.

    Key Indicators:HbO, HbR, and HbT concentration changes during a 0-40 sec task window. 3D topological maps (HbO beta values). Activation levels at rest. Functional connectivity (HbO).
11. Gait Analysis Laboratory

    A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for gait analysis. This non-invasive system captures:

    Spatiotemporal Parameters: Step time, frequency, speed, stride length/width, and symmetry Kinematic Parameters: Joint angles (pelvis, hip, knee), motion curves, ground reaction forces, and joint torques
12. Gut Microbiota and Blood Metabolomics Mid-portion fecal samples and 5 mL blood samples will be collected. Fecal samples will undergo non-targeted microbiome analysis at Novogene, while blood samples will be analyzed at Biotree Bioscience for metabolomic profiling, including appetite-related hormones such as ghrelin and PYY.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 20 to 70 years old;
* Rehabilitation patients with stroke or motor injuries;

Exclusion Criteria:

* Loss of autonomous mobility;
* Loss of consciousness;
* Individuals with metallic implants (e.g., pacemakers);
* Severe metabolic diseases (e.g., diabetes, other hereditary metabolic disorders);
* Patients with claustrophobia;
* Individuals with anorexia nervosa;
* Women in the preconception period, pregnancy, or lactation;
* Uremic patients;
* Inability to lie flat for one hour.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 20 to 70 years, both male and female, who are recovering from stroke or motor injuries are eligible for this study; however, those with the following conditions are not permitted to participate: pregnancy, pre-pregnancy period, lactation, loss of consciousness or mobility, severe metabolic diseases (such as diabetes, other hereditary metabolic disorders, etc.), psychogenic anorexia, uremia, and inability to lie flat for one hour. Additionally, individuals with contraindications for magnetic resonance imaging (MRI) are excluded from this trial; these include a history of pacemaker implantation, presence of metallic implants in the body, and claustrophobia. This criterion ensures that all participants meet the necessary health and safety requirements for the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Height | Height will be measured on the first day after volunteers are enrolled.
  Measured by seca 217 stable stadiometer. Subjects wearing no shoes.
Resting Energy Expenditure (REE) | The measurement of REE will be completed within fifteen days after the volunteers are enrolled.
  REE will be measured via indirect calorimetry using a respiratory hood system (Cosmed). Participants will report to the laboratory after an overnight fast, lie supine on a flat bed, and have the hood placed over their head. Oxygen consumption and carbon dioxide production will be recorded for 40 minutes, with the final 10 minutes used for analysis. The system will be quality-checked regularly using a turbine test, and monthly validation will be conducted via an alcohol combustion test.
Total Energy Expenditure (TEE) | The measurement of TEE will be completed within fifteen days after the volunteers are enrolled.
  TEE will be assessed using two complementary methods:
  Doubly Labeled Water (DLW) Method: Urine samples from the DLW subset will be stored at -20 °C and shipped on dry ice to Shenzhen Institutes of Advanced Technology, Chinese Academy of Sciences. Isotope ratios will be analyzed using a Liquid Water Isotope Analyzer (ABB). CO₂ production will be calculated using the latest equation from Speakman et al. (2021, Cell Reports Medicine), and TEE will be estimated using the Weir equation.
  Metabolic Chamber: TEE will also be measured using a whole-body metabolic chamber (Maastricht Instruments, Netherlands), which continuously tracks oxygen consumption and carbon dioxide production. Participants will remain in the chamber for 48 hours, engaging in routine daily activities. Data from the second day will be analyzed to estimate TEE.
Physical Activity Level | GT3X will be worn by the volunteers on the first day of enrollment and continue for fifteen days.
  During the measurement period, all participants will be required to wear a three-axis accelerometer (Actigraph GT3XP-BTLE, USA) for 15 days, covering 24 hours a day, including sleep. Participants can remove the accelerometer only when showering, bathing, swimming, or engaging in other water activities. This device will provide multiple parameters of physical activity levels, including raw acceleration data, activity counts, and vector magnitudes. Raw acceleration data captures subtle changes in individual movements, activity counts measure the intensity of physical activity over specific time periods, and vector magnitudes integrate acceleration information from all directions. These three indicators were used to comprehensively evaluate participants' physical activity levels.
Fat mass | Fat mass will be completed within fifteen days after the volunteers are enrolled.
  Fat mass will be measured by Magnetic Resonance Imaging (Philips Multiva 1.5T ).
Mental Health Assessment | Mental health assessment will be completed within fifteen days after the volunteers are enrolled.
  The Symptom Checklist-90 (SCL-90) will be used to evaluate psychological well-being. This tool measures ten dimensions: somatization, obsessive-compulsive traits, interpersonal sensitivity, depression, anxiety, hostility, phobia, paranoid ideation, psychosis, and additional symptoms. Scores for each dimension and overall symptom severity will be calculated.
Cognitive Function Assessment | Cognitive function assessment will be completed within fifteen days after the volunteers are enrolled.
  Cognitive performance will be evaluated using:
  Mini-Mental State Examination (MMSE): Assesses orientation, memory, attention, language, and visuospatial function. Scores of 25-30 indicate normal function; 20-24 mild, 10-19 moderate, and <10 severe cognitive impairment.
Fat free mass | Fat free mass will be completed within fifteen days after the volunteers are enrolled.
  Fat free mass will be measured by Bioimpedance Analysis (Tanita, Philips Multiva 1.5T).
Body weight | Body weight will be measured on the first day after volunteers are enrolled.
  Subjects will be asked to fast overnight and weight will be measured using a calibrated Seca body weight scale first thing in the morning on subjects wearing light clothes and no shoes. .
Cognitive Function Assessment | Cognitive function assessment will be completed within fifteen days after the volunteers are enrolled.
  Cognitive performance will be evaluated using:
  Montreal Cognitive Assessment (MoCA): Screens for impairment across eight cognitive domains. A score ≥26 is considered normal.
Bone mass | Bone mass will be completed within fifteen days after the volunteers are enrolled.
  Bone mass will be measured by DXA (HOLOGIC Horizon Wi，America）
Hunger Sensation | Hunger sensation assessment will be completed within fifteen days after the volunteers are enrolled.
  After enjoying a standardized lunch, designed according to the energy distribution recommendations and formula method outlined in the Chinese Dietary Guidelines, participants will receive a test meal five hours later. The meal, with its packaging removed, includes preset macro-nutrient and energy levels, allowing participants to determine their intake. Hunger sensation will be assessed using a VAS (Visual Analog Scale) for hunger.
PYY | PYY will be measured within fifteen days after the volunteers are enrolled.
  After enjoying a standardized lunch, designed according to the energy distribution recommendations and formula method outlined in the Chinese Dietary Guidelines, participants will receive a test meal five hours later. The meal, which has been removed from its packaging, includes preset macronutrient and energy levels, allowing participants to determine their intake. Blood samples are collected at 15,30, and 60 minutes before dinner, after dinner, and again before bedtime, with each sample being 2ml (a total of four times, with a permanent indwelling needle). PYY is detected through these blood samples.
Ghrelin | Ghrelin will be measured within fifteen days after the volunteers are enrolled.
  After enjoying a standardized lunch, designed according to the energy distribution recommendations and formula method outlined in the Chinese Dietary Guidelines, participants will receive a test meal five hours later. The meal, which has been removed from its packaging, includes preset macronutrient and energy levels, allowing participants to determine their intake. Blood samples are collected at 15,30, and 60 minutes before dinner, after dinner, and again before bedtime, with each sample being 2ml (a total of four times, with a permanent indwelling needle). Ghrelin is detected through these blood samples.
Total Sleep Duration | Total sleep duration will be completed within fifteen days after the volunteers are enrolled.
  Total sleep duration will be monitored using the Xinxiaoyouhu Pro AI Precision Health Management System.
Sleep Efficiency | Sleep efficiency will be completed within fifteen days after the volunteers are enrolled.
  Sleep efficiency will be monitored using the Xinxiaoyouhu Pro AI Precision Health Management System.
Sleep Cycle Durations | Sleep cycle durations will be completed within fifteen days after the volunteers are enrolled.
  Sleep cycle durations will be monitored using the Xinxiaoyouhu Pro AI Precision Health Management System.
Heart Rate During Sleep | Heart rate during sleep will be completed within fifteen days after the volunteers are enrolled.
  Heart rate during sleep will be monitored using the Xinxiaoyouhu Pro AI Precision Health Management System.
Respiratory Patterns During Sleep | Respiratory patterns during sleep will be completed within fifteen days after the volunteers are enrolled.
  Respiratory patterns during sleep will be monitored using the Xinxiaoyouhu Pro AI Precision Health Management System.
Step Time | Step time will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for step time.
Step Frequency | Step frequency will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for step frequency.
Step Speed | Step speed will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for step speed.
Stride Length | Stride length will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for stride length.
Bilateral Gait Symmetry | Bilateral gait symmetry will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for bilateral gait symmetry.
Pelvic, Hip and Knee Joint Angle Parameters | Pelvic, hip and knee joint Angle parameters will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for pelvic, hip and knee joint angle parameters.
Joint Torque | Joint torque will be completed within fifteen days after the volunteers are enrolled.
  A 3D markerless motion capture system (Xiangneng-Dongxi) will be used for joint torque.
Non-Targeted Microbiome Detection Of Stool Samples | The retention of stool samples for non-targeted microbiome detection will be completed within 15 days after the enrollment of volunteers, and the sample analysis will be completed before November 1, 2025.
  Non-targeted microbiome studies are a comprehensive and unbiased approach to studying microbial communities. This method uses high-throughput sequencing or mass spectrometry to analyze the genomes (metagenomics) or metabolites (metabolomics) of all microorganisms in a sample, without preconceived targets. Since this study does not have a specific target microorganism, we will collect approximately 10ml of midstream fecal samples from participants for the detection of all microorganisms' genomes (metagenomics) or metabolites (metabolomics).
Non-Invasive Brain Function Monitoring | Non-invasive brain function monitoring will be completed within fifteen days after the volunteers are enrolled.
  Functional Near-Infrared Spectroscopy (fNIRS) will be used to assess brain activity by measuring changes in oxyhemoglobin and deoxyhemoglobin concentrations. We may use the BS2000 near-infrared imaging system for this purpose.
  Assessment Areas: Prefrontal cortex, motor cortex, frontal pole, dorsolateral prefrontal cortex, primary motor/somatosensory cortex, premotor and supplementary motor cortex-on both healthy and affected sides.
  Key Indicators:HbO, HbR, and HbT concentration changes during a 0-40 sec task window. 3D topological maps (HbO beta values). Activation levels at rest. Functional connectivity (HbO).
Cerebral Oxyhemoglobin Concentration | Cerebral oxyhemoglobin concentrationn will be completed within fifteen days after the volunteers are enrolled.
  Functional Near-Infrared Spectroscopy (fNIRS) will be used to measured cerebral oxyhemoglobin concentration.
Cerebral Deoxyhemoglobin Concentration | Cerebral deoxyhemoglobin concentration will be completed within fifteen days after the volunteers are enrolled.
  Functional Near-Infrared Spectroscopy (fNIRS) will be used to measured cerebral deoxygenated concentration.
Total Hemoglobin Concentration In Cerebral Vasculature | Total hemoglobin concentration in cerebral vasculature will be completed within fifteen days after the volunteers are enrolled.
  Functional Near-Infrared Spectroscopy (fNIRS) will be used to measured total hemoglobin concentration in cerebral vasculature

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Zhang, PhD, Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences; John R Speakman, PhD, Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Guangdong Jianxiang Hospital Group, Foshan, Guangdong, China

REFERENCES:
- [Background] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301